CLINICAL TRIAL: NCT06808984
Title: A Phase 2, Randomized, Double-blind, Three-Arm, Placebo-controlled, Multicenter Study Assessing the Efficacy, Safety and Tolerability of Orally Administered BMS-986368, a FAAH/MAGL Inhibitor, for the Treatment of Agitation in Participants With Alzheimer's Disease (BALANCE-AAD-1)
Brief Title: Study to Evaluate the Efficacy, Safety, and Tolerability of BMS-986368, for the Treatment of Agitation in Participants With Alzheimer's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IM045-P06; U1111-1313-8997 (Other: WHO)
Record Dates: First submitted 2025-01-24; First posted 2025-02-05 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Agitation; Alzheimer Disease
MeSH Terms: conditions — Psychomotor Agitation; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BMS-986368 Dose 1 (Experimental)
  Interventions: Drug: BMS-986368
- BMS-986368 Dose 2 (Experimental)
  Interventions: Drug: BMS-986368
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMS-986368 — Specified dose on specified days
  Other Names: CC-97489
  Arms: BMS-986368 Dose 1; BMS-986368 Dose 2
Drug: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
This is a study to evaluate the efficacy, safety, and tolerability of BMS-986368, a FAAH/MAGL inhibitor, for the treatment of agitation in participants with Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of Alzheimer's disease with biomarker confirmation meeting the 2024 Revised criteria for diagnosis and staging of AD: Alzheimer's Association Workgroup.
* The diagnosis of agitation must meet the International Psychogeriatric Association (IPA) definition of agitation.
* History of agitation with onset at least four weeks prior to Screening
* MMSE-1 score < 21
* NPI-NH agitation/aggression sub-score ≥ 4.
* Stable living environment for at least 6 weeks prior to Screening. Participants are eligible if they are in nursing homes, assisted living facilities, or living at home and have an identified study partner (caregiver).
* Capable of self-locomotion (alone or with the aid of an assistive device); wheelchairs and other mobility aids are acceptable.

Exclusion Criteria:

* Clinically significant delusions/hallucinations requiring hospitalization.
* History of bipolar disorder, schizophrenia, or schizoaffective disorder.
* History of major depressive episode with psychotic features during the 12 months prior to Screening.
* History of delirium within 30 days of Screening.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2027-11-26 (Estimated); Study Completion 2028-01-07 (Estimated)

PRIMARY OUTCOMES:
Change in Cohen-Mansfield Agitation Inventory (CMAI) total score from baseline | Up to Week 8
  The CMAI is a scale administered by qualified rater based on caregiver's input on 29 items that assess the frequency of manifestations of agitated behaviors in older adults. Each item is rated on a 7-point scale: 1 = "never", 2 = "less than once a week", 3 = "once or twice a week", 4 = "several times a week", 5 = "once or twice a day", 6 = "several times a day" and 7 = "several times per hour." Ratings pertain to the period of time over the previous 2 weeks preceding administration of the CMAI. CMAI total scores range from 29 to 203.

SECONDARY OUTCOMES:
Change in Clinical Global Impression-Severity (CGI-S) | Up to Week 8
Change in CMAI-International Psychogeriatric Association (CMAI-IPA) Total Score | Up to Week 8
CMAI sub-score change in Aggressive Behaviors | Up to Week 8
CMAI sub-score change in Physically Non-aggressive Behaviors | Up to Week 8
CMAI sub-score change in Verbally Agitated Behaviors | Up to Week 8
Change in Neuropsychiatric Inventory Nursing Home Version (NPI-NH) Total Score | Up to Week 8
Change in NPI-NH Agitation/Aggression Domain Score | Up to Week 8
Change in NPI-NH Occupational Disruptiveness for Agitation/aggression Domain | Up to Week 8
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Up to Day 28 After Last Dose
Number of Participants with Serious Adverse Events (SAEs) | Up to Day 28 After Last Dose
Number of Participants with Adverse Events (AEs) | Up to Day 28 After Last Dose
Number of Participants with Clinically Significant Laboratory Abnormalities | Up to 28 Days After Last Dose
Change in Suicidal Ideation Assessed by Sheehan-Suicidality Tracking Scale (S-STS) | Up to Day 28 After Last Dose
Change in Behaviour Assessed by Sheehan-Suicidality Tracking Scale (S-STS) | Up to Day 28 After Last Dose
Abuse Potential Assessed by the Cannabis Withdrawal Scale (CWS) | Up to Day 21 After Last Dose
Withdrawal Symptoms Assessed by the Cannabis Withdrawal Scale (CWS) | Up to Day 21 After Last Dose
Plasma Concentrations of BMS-986368 | Up to Week 14

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (52):
- United States (52):
  - Local Institution - 0046, Homewood, Alabama
  - University of Alabama - Huntsville Regional Medical Campus, Huntsville, Alabama
  - NoesisPharma, Phoenix, Arizona
  - Local Institution - 0040, Scottsdale, Arizona
  - Local Institution - 0017, Anaheim, California
  - Inland Psychiatric Medical Group, Inc, Chino, California
  - Kaizen Brain Center, La Jolla, California
  - University of California San Diego - La Jolla, La Jolla, California
  - Shreenath Clinical Service - Lakewood, Lakewood, California
  - Accellacare - Sherman Oaks, Sherman Oaks, California
  - Next Level Clinical Trials, West Covina, California
  - Alliance Clinical -West Hills, West Hills, California
  - Local Institution - 0066, Aurora, Colorado
  - Local Institution - 0053, Washington D.C., District of Columbia
  - Arrow Clinical Trials, Daytona Beach, Florida
  - ClinCloud, Maitland, Florida
  - Local Institution - 0007, Maitland, Florida
  - Local Institution - 0022, Miami, Florida
  - Ocean Blue Medical Research Center, Miami, Florida
  - Local Institution - 0001, Tampa, Florida
  - Charter Research - Lady Lake, The Villages, Florida
  - Advanced Discovery Research, Atlanta, Georgia
  - CenExel iResearch, LLC, Decatur, Georgia
  - CenExel iResearch, LLC, Savannah, Georgia
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Local Institution - 0011, Marrero, Louisiana
  - Local Institution - 0051, South Dartmouth, Massachusetts
  - Local Institution - 0061, Missoula, Montana
  - Be Well Clinical Studies - Omaha, Omaha, Nebraska
  - Oasis Clinical Trials, Las Vegas, Nevada
  - Local Institution - 0059, Livingston, New Jersey
  - University at Buffalo - UBMD Neurology, Buffalo, New York
  - The Feinstein Institute for Medical Research, Manhasset, New York
  - Mid Hudson Medical Research, New Windsor, New York
  - Hawthorne Health - Super Health Staten Island, Staten Island, New York
  - Research Central LLC (DBA Ichor Research), Syracuse, New York
  - New Hope Clinical Research, Charlotte, North Carolina
  - Local Institution - 0063, Raleigh, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Local Institution - 0058, Philadelphia, Pennsylvania
  - K2 Medical Research - East Providence, East Providence, Rhode Island
  - Local Institution - 0031, Chattanooga, Tennessee
  - Neurology Clinic, P.C., Cordova, Tennessee
  - Vanderbilt University Medical Center- Village, Nashville, Tennessee
  - Pinnacle Clinical Research, Austin, Texas
  - Horizon Clinical Research Center - Houston, Cypress, Texas
  - ANESC Research, El Paso, Texas
  - North Pointe Psychiatry - Flower Mound, Flower Mound, Texas
  - Local Institution - 0020, Houston, Texas
  - Local Institution - 0065, Plano, Texas
  - Be Well Clinical Studies, Round Rock, Texas
  - Boeson Research - Provo, Provo, Utah

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06808984.html